CLINICAL TRIAL: NCT02124135
Title: Eat Out With KP: A Pilot to Improve the Impact of Dietary Advice for Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Kristina Lewis, Assistant Investigator, Kaiser Permanente
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00004774
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Obesity
Keywords: Nutrition
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clinic-based counseling (Active Comparator): Participants in this arm will receive 1 baseline phone call with the registered dietitian to get preliminary dietary counseling tailored to their family's needs. They will then have 3 sessions in-person in a group setting with another family and the registered dietitian where a set dietary curriculum geared at promoting weight loss and/or maintenance of a healthy weight will be emphasized. All in-person visits will take place in the clinic setting.
  Interventions: Behavioral: Diet/Nutrition Education
- Restaurant-based counseling (Experimental): Participants in this arm will receive 1 baseline phone call with the registered dietitian to get preliminary dietary counseling tailored to their family's needs. They will then have 3 sessions in-person in a group setting with another family and the registered dietitian where a set dietary curriculum geared at promoting weight loss and/or maintenance of a healthy weight will be emphasized. All in-person visits will take place in a restaurant, while dining.
  Interventions: Behavioral: Diet/Nutrition Education

INTERVENTIONS:
Behavioral: Diet/Nutrition Education — As described elsewhere, all participants will receive 1 phone call and 3 in person sessions with the registered dietitian.
  Participants in the "clinic" arm will receive the education intervention in the clinic.
  Participants in the "restaurant" arm will receive the education intervention while dining in a restaurant.

SUMMARY:
Dietary counseling at the point of purchase could improve patient adherence to dietary advice and downstream health outcomes. The aim of our pilot is to test the efficacy of a novel delivery system for dietary advice. We will study the effect of relocating family weight management counseling sessions into restaurants, where registered dieticians and patients will conduct scheduled group visits while enjoying a meal together. As with office-based visits, our goal is for members and their families to learn how to select food options based on their unique health needs, budgetary concerns, and time constraints. In contrast to a traditional counseling visit, however, co-dining with a dietitian will give members a hands-on experience designed to enhance their learning and improve adherence. The proposed study would build on an existing pilot of a similar program, the "KP Personal Shopper", where dietitian visits were conducted with individuals either in the clinic setting or while shopping in a grocery store.

We will compare the new "Eat Out with Kaiser" approach to the current standard of clinic-based dietary and lifestyle counseling for weight management among 40 families affected by obesity, with the following outcomes in mind:

1. Change in dietary measures
2. Nutritional knowledge of families
3. Participant self-efficacy and confidence in food purchasing decisions
4. Participant and dietician perception of visit

We hypothesize that, compared to clinic-based visits, our "Eat Out with Kaiser" visits will result in more favorable perception of the visit by both dietitian and participant, higher nutritional knowledge scores, higher self-efficacy and confidence of patients around food decisions, and larger improvements in diet components.

DETAILED DESCRIPTION:
Dietary counseling at the point of purchase could improve patient adherence to dietary advice and downstream health outcomes. The aim of our pilot is to test the efficacy of a novel delivery system for dietary advice. We will study the effect of relocating family weight management counseling sessions into restaurants, where registered dieticians and patients will conduct scheduled group visits while enjoying a meal together. As with office-based visits, our goal is for members and their families to learn how to select food options based on their unique health needs, budgetary concerns, and time constraints. In contrast to a traditional counseling visit, however, co-dining with a dietitian will give members a hands-on experience designed to enhance their learning and improve adherence. The proposed study would build on an existing pilot of a similar program, the "KP Personal Shopper", where dietitian visits were conducted with individuals either in the clinic setting or while shopping in a grocery store.

Our study population will come from a local employer group, and we will use the electronic medical record to identify families where at least one child and one parent are affected by obesity. Assuming families are interested and meet eligibility criteria, they will be enrolled in the study.

Our study design is a randomized trial, where randomization occurs at the unit of the family. 45 families will be randomized into one of two arms. All families will receive a baseline 30 minute phone call with the dietitian, followed by three in-person group visits. Those in the intervention (Eat Out) arm will have their in-person visits conducted during mealtimes at a restaurant. Those in the control (clinic) arm will have their in-person visits conducted in a classroom at a Kaiser medical office building.

We will compare the new "Eat Out with Kaiser" approach to the current standard of clinic-based dietary and lifestyle counseling for weight management among 40 families affected by obesity, with the following outcomes in mind:

1. Change in dietary measures including - Fruit and Vegetable Intake, Whole Grain Intake, Saturated Fat Intake and Added Sugars.
2. Nutritional knowledge of families
3. Participant self-efficacy and confidence in food purchasing decisions - all family members
4. Participant and dietician perception of visit type (attendance, feasibility, effectiveness, e.g.)

We hypothesize that, compared to clinic-based visits, our "Eat Out with Kaiser" visits will result in more favorable perception of the visit by both dietitian and participant, higher nutritional knowledge scores, higher self-efficacy and confidence of patients around food decisions, and larger improvements in diet components.

ELIGIBILITY:
Inclusion Criteria:

* adult member of Kaiser Georgia, in a specific employer group
* families in which at least one parent and one child are obese
* family with 2 or fewer children all between 8-13 years of age
* no-show rate for clinic visits <10%
* adult is 18-64 years of age

Ages: 8 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 94 (Actual)
Dates: Start 2014-05; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in Fruit and Vegetable Intake | 3 months
  Will be measured in one parent and one child per enrolled family using the Block food screeners for adults and children.
Change in Whole Grain Intake | 3 months
  Will be measured in one parent and one child per enrolled family using the Block food screeners for adults and children.
Change in Saturated Fat Intake | 3 months
  Will be measured in one parent and one child per enrolled family using the Block food screeners for adults and children.
Change in Added Sugars Intake | 3 months
  Will be measured in one parent and one child per enrolled family using the Block food screeners for adults and children.

SECONDARY OUTCOMES:
Change in Nutritional Knowledge of Families | 3 months
  Will be assessed using a modified version of previously validated nutritional knowledge from the UK. Total possible score of 65 points. Covers topics such as recommendations from experts, types of fat, foods high in sodium, added sugar, fiber and fat.
Self-efficacy around food purchasing and dietary decisions | 3 months
  Will be assessed using a series of questions about how confident a participant feels about his / her ability to change food and dietary behaviors in the near future. Paper survey to be administered to one adult per participating family.

CONTACTS AND LOCATIONS:
Overall Officials: Kristina H Lewis, MD MPH SM, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Center for Health Research, Southeast, Atlanta, Georgia, United States